CLINICAL TRIAL: NCT06792955
Title: A Single-center, Single-dose, Randomized, Open-label, Single-period, Parallel Bioequivalence Study of HRS9531 Injection Solution in Multi-dose Pens and Single-dose Pens in Overweight/Obese Subjects
Brief Title: The Evaluation of Bioequivalence Between a Single-dose Pen and a Multi-dose Pen of HRS9531 Injection Solution
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Fujian Shengdi Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HRS9531-108
Record Dates: First submitted 2025-01-20; First posted 2025-01-27 (Actual); Last update posted 2025-06-12 (Actual); Status verified 2025-06

CONDITIONS: Overweight/Obesity
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment group R (Experimental): Multi-dose pen of HRS9531 injection solution.
  Interventions: Drug: HRS9531 injection
- Treatment group T (Experimental): Single-dose pen of HRS9531 injection solution.
  Interventions: Drug: HRS9531 injection

INTERVENTIONS:
Drug: HRS9531 injection — Multi-dose pen of HRS9531 injection solution.
  Arms: Treatment group R
Drug: HRS9531 injection — Single-dose pen of HRS9531 injection solution.
  Arms: Treatment group T

SUMMARY:
The study is being conducted to evaluate the bioequivalence between a single-dose pen and a multi-dose pen of HRS9531 injection solution.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must provide informed consent prior to the trial, demonstrating a full understanding of the trial's content, procedures and potential adverse reactions, and willingly sign a written informed consent form. They must also be willing and capable of adhering to the trial protocol to complete the study.
2. On the day of signing the informed consent form, the subjects must be overweight/obese males or females aged 18 to 45 years inclusive of the boundary values.
3. From the time of signing the informed consent form until two months after the last drug administration, subjects must have no plans for conception (for both male and female subjects) and must voluntarily adopt effective contraceptive measures. They must also have no plans to donate eggs/sperm. Female subjects of reproductive potential must have a negative pregnancy test.

Exclusion Criteria:

1. Subjects with a history of primary diseases in major organs, including but not limited to the nervous system, mental system, cardiovascular system, digestive system, respiratory system, urinary system, endocrine system, hematopoietic system and immune system, as judged by the investigator to be unsuitable for participation in this trial.
2. Subjects with a history of significant gastric emptying abnormalities or factors affecting gastric emptying, or clinically significant gastrointestinal diseases, or those who have undergone gastrointestinal surgery (excluding polypectomy, appendectomy and hemorrhoidectomy).
3. Subjects who have undergone any surgery within 6 months prior to dosing, or those planning to undergo surgical procedures during the study period.
4. Subjects who have experienced blood loss or donated blood ≥400 mL within 3 months prior to dosing or ≥200 mL within 1 month prior to dosing, or those who have received a blood transfusion within 3 months prior to dosing.
5. Subjects who are positive for Hepatitis B surface antigen (HBsAg), Hepatitis C virus antibody (HCVAb), Human Immunodeficiency Virus (HIV) antibody or Treponema pallidum-specific antibody.
6. Subjects with a history of drug use or abuse within 1 year prior to dosing, or those with a positive drug screen.
7. Subjects who are heavy users of alcohol and tobacco (consuming an average of ≥14 units of alcohol per week for the 6 months prior to screening: 1 unit = 285 mL of beer, or 25 mL of spirits, or 100 mL of wine; smoking ≥5 cigarettes per day on average) and who are unable to abstain as required by the protocol during the trial; those with a positive alcohol screen; those with a positive cotinine screen.
8. Subjects who have consumed foods or beverages containing methylxanthines (such as tea, coffee, cola, chocolate, energy drinks) or alcohol, or have engaged in vigorous exercise within 72 hours prior to the first use of the trial medication.
9. Nursing women.
10. Subjects with a history of fainting at the sight of needles or blood, difficulty in drawing blood, or inability to tolerate venous blood collection.
11. Subjects with special dietary habits that the investigator deems unsuitable for participation, or those who cannot follow the dietary requirements of the trial during the study period.
12. Subjects who have received or plan to receive live (attenuated) vaccines within 1 month prior to dosing or during the trial (except for influenza vaccines).
13. Subjects whom the investigator deems to have any other factors that make them unsuitable for this trial, or those who withdraw from the study for personal reasons.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2025-02-11 (Actual); Primary Completion 2025-06-06 (Actual); Study Completion 2025-06-06 (Actual)

PRIMARY OUTCOMES:
The maximum plasma concentration (Cmax) | Post-dose at day 1 to day 43.
Area under the concentration curve from time 0 to the last quantifiable concentration (AUClast) | Post-dose at day 1 to day 43.
Area under the concentration curve from time 0 to extrapolated infinite time (AUCinf) | Post-dose at day 1 to day 43.

SECONDARY OUTCOMES:
Time to maximum plasma concentration (Tmax) | Post-dose at day 1 to day 43.
Terminal half-life (t1/2) | Post-dose at day 1 to day 43.
Apparent clearance (CL/F) | Post-dose at day 1 to day 43.
Apparent volume of distribution (Vz/F) | Post-dose at day 1 to day 43.
Incidence and severity of adverse events (AEs) | Screening period up to day 43.

CONTACTS AND LOCATIONS:
Locations (1):
- Central Hospital Affiliated To Shandong First Medical University, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: Undecided